CLINICAL TRIAL: NCT04768517
Title: Risk of Hepatitis C Virus Reinfection in Human Immunodeficiency Virus and Hepatitis C Virus Coinfected Patients Achieving Sustained Virologic Response by Antiviral Therapy
Brief Title: HCV Reinfection in in HIV/HCV-coinfected Patients Achieving SVR by Antiviral Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202012260RIND
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Hepatitis C Virus Infection; Hepatitis C Virus Infection, Response to Therapy of; Human Immunodeficiency Virus (HIV) Coinfection
Keywords: Hepatitis C virus; Human immunodeficiency virus; Sustained virologic response; Reinfection
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome; Coinfection; Reinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic hepatitis C virus (HCV) infection remains a health burden in people living with human immunodeficiency virus (HIV). Interferon (IFN)-based therapy is the treatment of choice for HCV infection for HIV coinfected patients in earlier years. However, the treatment responses are far from ideal and the treatment-emergent adverse events (AEs) are frequently encountered. Based on the excellent efficacy and safety, IFN-free direct acting antivirals (DAAs) have been the mainstay of therapy for HCV. Furthermore, the world health organization (WHO) has set the goal of global HCV elimination by 2030. The microelimination of HCV among HIV/HCV-coinfected patients is also listed as the prioritized target by WHO. Although the overall treatment response has improved dramatically during the past 5-10 years, several studies have indicated the HIV/HCV-coinfected patients had high risks of reinfection following successful antiviral treatment. The risk of HCV reinfection was reported to be 24.6% among HIV-positive men who have sex with men (MSM) in Austria, German, France and the United Kingdom who attained sustained virologic response (SVR) by IFN-based therapy. Two recent studies from Canada showed that the incidence of HCV reinfection in HIV-positive patients was higher that HIV-negative patients (3.44 vs. 1.13 per 100 person-year; 2.56 vs. 1.12 per 100 person-year). In Taiwan, 14.1% of the HIV-positive patients had HCV reinfection following treatment-induced or spontaneous viral clearance, resulting an incidence of 8.2 per 100 person-year with a total of 218.3 person-years of follow-up for these patients.

Because data regarding to the HCV reinfection in HIV-positive patients are still limited, where a more comprehensive assessment of HCV reinfection is important based on the perspectives of HCV microelimination among HIV-positive patients in Taiwan, the investigators thus aim to conduct a long-term, large-scale cohort study to assess the risk of HCV reinfection in HIV-positive patients achieving SVR after IFN-based or IFN-free therapies, and to assess the factors associated with different risks of reinfection in these patients.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection remains a health burden in people living with human immunodeficiency virus (HIV). Compared to the midpoint prevalence rate of HCV coinfection to be 2.4% in the general HIV-positive population, the prevalence rates are higher among bisexual men (4.0%), gay men (6.4%), and people who inject drugs (PWIDs) (82.4%). Following the widespread use of antiretroviral therapy (ART) for HIV which improves the health outcome by reducing the acquired immunodeficiency syndrome (AIDS)-related deaths, the liver-related death has become a frequent cause of non-AIDS-related deaths in HIV-positive population. If HCV is left untreated, the HIV/HCV-coinfected patients may have higher risks of developing hepatic decompensation or hepatocellular carcinoma (HCC) than HCV-monoinfected patients due to the accelerated progression of hepatic fibrosis.

Interferon (IFN)-based therapy is the treatment of choice for HCV infection for HIV coinfected patients in earlier years. However, the treatment responses are far from ideal and the treatment-emergent adverse events (AEs) are frequently encountered. Based on the excellent efficacy and safety, IFN-free direct acting antivirals (DAAs) have been the mainstay of therapy for HCV. Furthermore, the world health organization (WHO) has set the goal of global HCV elimination by 2030. The microelimination of HCV among HIV/HCV-coinfected patients is also listed as the prioritized target by WHO.

Although the overall treatment response has improved dramatically during the past 5-10 years, several studies have indicated the HIV/HCV-coinfected patients had high risks of reinfection following successful antiviral treatment. The risk of HCV reinfection was reported to be 24.6% among HIV-positive men who have sex with men (MSM) in Austria, German, France and the United Kingdom who attained sustained virologic response (SVR) by IFN-based therapy. Two recent studies from Canada showed that the incidence of HCV reinfection in HIV-positive patients was higher that HIV-negative patients (3.44 vs. 1.13 per 100 person-year; 2.56 vs. 1.12 per 100 person-year). In Taiwan, 14.1% of the HIV-positive patients had HCV reinfection following treatment-induced or spontaneous viral clearance, resulting an incidence of 8.2 per 100 person-year with a total of 218.3 person-years of follow-up for these patients.

Because data regarding to the HCV reinfection in HIV-positive patients are still limited, where a more comprehensive assessment of HCV reinfection is important based on the perspectives of HCV microelimination among HIV-positive patients in Taiwan, the investigators thus aim to conduct a long-term, large-scale cohort study to assess the risk of HCV reinfection in HIV-positive patients achieving SVR after IFN-based or IFN-free therapies, and to assess the factors associated with different risks of reinfection in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age old than 20 years old
* Patients with human immunodeficiency virus coinfection (HIV) during IFN-based or IFN-free antiviral therapy for hepatitis C virus (HCV) infection
* Patients achieving SVR, defined as undetectable serum HCV RNA at week 12 off-therapy

Exclusion Criteria:

* Poor access to sites for venipuncture

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV/HCV-coinfected patients who undergo antiviral therapy for hepatitis C virus infection and who achieve sustained virologic response
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative reinfection rate | Through study completion, an average of 3 years
  Time-dependent accumulative proportion of participants with evidence of resurgence of HCV viremia from the time point of viral clearance after antiviral therapy to the time point of last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Principal Investigator — National Taiwan University Hospital
Locations (7):
- Taiwan (7):
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei City Hospital, Ren-Ai Branch, Taipei
  - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital, Taipei